CLINICAL TRIAL: NCT03026959
Title: The Role of Mindfulness Skills Training in Maternal Mental Health: A Randomized Controlled Trial
Brief Title: Mindfulness and Maternal Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Dwight Mazmanian, Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 083 16-17
Record Dates: First submitted 2016-12-01; First posted 2017-01-20 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Group (Experimental): Participants assigned to the mindfulness group will attend four weekly sessions that are each 1.5 hours in length. The sessions will follow the structure described by Short, Mazmanian, Ozen, & Bédard (2015). The structure is designed to first enhance learners' foundation skills in mindfulness and progresses into teaching learners more advanced mindfulness skills.
  Interventions: Behavioral: Mindfulness
- Social (control) Group (No Intervention): Participants assigned to the social group will also attend four weekly sessions that are each 1.5 hours in length. Each session will have participants focus on a creative tasks while permitting task related discussion. In this way the format is designed to parallel the mindfulness group, where participants engage in a new activity each week and have an opportunity to discuss the activities with the group without engaging in any formal intervention.

INTERVENTIONS:
Behavioral: Mindfulness — The mindfulness intervention follows the structure described by Short, Mazmanian, Ozen, & Bédard, (2015).
  Arms: Mindfulness Group

SUMMARY:
There is preliminary empirical support for the use of mindfulness interventions during the perinatal period; suggesting that mindfulness training may be an effective treatment approach for reducing depression and anxiety symptoms during pregnancy and reducing anxiety, stress, and psychological distress during the postpartum period. To extend on these findings, the purpose of this research is to evaluate the effectiveness of a brief mindfulness-based program in protecting maternal mental health and well-being using a randomized controlled trial.

DETAILED DESCRIPTION:
Based on the results reported in the existing literature that show that formal mindfulness-based practice is effective for improving mental health status and preventing depressive symptom relapse, this research aims to evaluate the effectiveness of a brief mindfulness-based program, offered during pregnancy, in reducing mothers' psychological symptoms during pregnancy and the postpartum period. A brief program has the advantage being more economical to facilitate compared to full-length programs and also requires a shorter commitment from pregnant women, who are also attempting to manage multiple other new and existing demands (e.g., obstetrics appointments, work).

As emerging research suggests that women are particularly vulnerable to increased depressive, anxious, obsessive, compulsive, and hypomanic symptoms during the perinatal period these are the main psychological symptoms that will be assessed. As well, perceived stress and psychological resiliency will also be assessed for in order to examine changes in these domains in relation to mindfulness engagement. Furthermore, as a reduction in maternal psychological symptoms has been reported to have implications for mother-infant bond, the mother's interpersonal functioning, and maternal quality of life, the investigators will also assess to see if there are corresponding changes in these domains related to mindfulness engagement.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, age 18 years and older, able and willing to attend the study site for the four group sessions.

Exclusion Criteria:

* presence of a current severe mental health condition or mental heath difficulties that would be better addressed through another form of therapy, active major medical illness including significant obstetric complications, inability to give informed consent, inability to speak or understand English, at high risk for delivery before reaching full term (38 weeks gestation), or previous completion of a structured mindfulness-based program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 12 weeks postpartum
Hospital Anxiety and Depression Scale - Anxiety Subscale | 12 weeks postpartum
Obsessive-Compulsive Inventory-Revised | 12 weeks postpartum
Altman Self-Rating Mania Scale | 12 weeks postpartum
Five Facet Mindfulness Questionnaire | 12 weeks postpartum

SECONDARY OUTCOMES:
Perceived Stress Scale | 12 weeks postpartum
Brief Resilience Scale | 12 weeks postpartum
Postpartum Bonding Questionnaire | 12 weeks postpartum
World Health Organization Quality of Life Scale | 12 weeks postpartum
Multidimensional Scale of Perceived Social Support | 12 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Mazmanian, Ph.D, Principal Investigator — Lakehead University
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedard M, Felteau M, Marshall S, Cullen N, Gibbons C, Dubois S, Maxwell H, Mazmanian D, Weaver B, Rees L, Gainer R, Klein R, Moustgaard A. Mindfulness-based cognitive therapy reduces symptoms of depression in people with a traumatic brain injury: results from a randomized controlled trial. J Head Trauma Rehabil. 2014 Jul-Aug;29(4):E13-22. doi: 10.1097/HTR.0b013e3182a615a0. PMID 24052092
- [Background] Davey HL, Tough SC, Adair CE, Benzies KM. Risk factors for sub-clinical and major postpartum depression among a community cohort of Canadian women. Matern Child Health J. 2011 Oct;15(7):866-75. doi: 10.1007/s10995-008-0314-8. Epub 2008 Feb 7. PMID 18256913
- [Background] Helmes E, Ward BG. Mindfulness-based cognitive therapy for anxiety symptoms in older adults in residential care. Aging Ment Health. 2017 Mar;21(3):272-278. doi: 10.1080/13607863.2015.1111862. Epub 2015 Nov 13. PMID 26565928
- [Background] O'Hara MW, Wisner KL. Perinatal mental illness: definition, description and aetiology. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):3-12. doi: 10.1016/j.bpobgyn.2013.09.002. Epub 2013 Oct 7. PMID 24140480
- [Background] Pope CJ, Sharma V, Mazmanian D. Recognition, diagnosis and treatment of postpartum bipolar depression. Expert Rev Neurother. 2014 Jan;14(1):19-28. doi: 10.1586/14737175.2014.846219. Epub 2013 Nov 26. PMID 24308278
- [Background] Russell EJ, Fawcett JM, Mazmanian D. Risk of obsessive-compulsive disorder in pregnant and postpartum women: a meta-analysis. J Clin Psychiatry. 2013 Apr;74(4):377-85. doi: 10.4088/JCP.12r07917. PMID 23656845
- [Background] Short MM, Mazmanian D, Ozen LJ, Bédard M. Four days of mindfulness meditation training for graduate students: A pilot study examining effects on mindfulness, self-regulation, and executive function. J Contemplative Inq. 2015; 2(1). http://journal.contemplativeinquiry.org/index.php/joci/article/view/13